CLINICAL TRIAL: NCT04413825
Title: Diagnostic Accuracy of Early Systolic Notching in Pulmonary Embolism
Brief Title: Early Systolic Notching in Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: Akdeniz University (Other); Ege University (Other); Antalya Training and Research Hospital (Other Government); Rize Üniversitesi (Other); Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Aslaner, Assos. Prof., Gazi University
Other Study IDs: Gazi U.
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous thromboembolism (VTE), clinically seen as deep vein thrombosis (DVT) or pulmonary embolism (PE), is the third most common acute cardiovascular syndrome after myocardial infarction and stroke. In a study conducted by critical care and emergency physicians, lung ultrasonography (US) for pleural infarction areas, lower extremity venous US in terms of DVT, and focused cardiac US in terms of right ventricular strain were demonstrated with different diagnostic values for PE. However, no ultrasonographic method alone has a high diagnostic value for PE alone in the literature. In a recent study, it is stated that a new cardiac finding (early systolic notch- ESN) has high sensitivity (92%) and specificity (99%) in massive and submassive emboli. However, the limited patient population and the exclusion of many patient groups limits the applicability of the study and its use in other patient groups. With this study, it was aimed to determine the diagnostic value of ESN finding within the emergency department conditions by keeping the patient population wider.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pulmonary CT angiography with suspicion of pulmonary embolism

Exclusion Criteria:

* Pregnant women,
* Patients under 18 years of age,
* Those who received thrombolytic therapy,
* Poor ultrasound imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented to the emergency department and underwent pulmonary CT angio imaging with suspicion of pulmonary embolism.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
To determine the diagnostic accuracy of the ESN finding | 6 months
  What is the diagnostic value of ESN finding in patients with PE diagnosed with pulmonary CT angio?

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Facaulty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided